CLINICAL TRIAL: NCT05766891
Title: Opioid-Sparing Effects of Nurse-Delivered Hypnosis During Breast Cancer Surgery
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rising Tide Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0959; NCI-2023-02059 (Other: NCI-CTRP Clinical Trials Registry); 5R01CA272565 (NIH); CCR-23-500 (Other Grant/Funding Number: Rising Tide Foundation for Clinical Cancer Research)
Record Dates: First submitted 2023-03-02; First posted 2023-03-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Participants will receive hypnosedation before and during surgery as well as local anesthesia and pain/nausea medications during surgery
  Interventions: Behavioral: Group 1
- Group 2 (Experimental): Participants will receive hypnosedation before surgery and standard general anesthesia during surgery.
  Interventions: Behavioral: Group 2
- Group 3 (Experimental): Participants will receive standard general anesthesia alone. You will not receive hypnosedation.
  Interventions: Behavioral: Group 3

INTERVENTIONS:
Behavioral: Group 1 — Participants will receive hypnosedation will be restarted after arriving in the operating room and will continue for the whole time of surgery
  Arms: Group 1
Behavioral: Group 2 — Participants will receive standard general anesthesia and medications to control your pain after arriving in the operating room
  Arms: Group 2
Behavioral: Group 3 — Participants will receive standard general anesthesia and medications during surgery to control your pain.
  Arms: Group 3

SUMMARY:
To hypnosedation alone given before and during surgery on reducing opioid use after surgery compared to standard general anesthesia given alone or with hypnosedation.

DETAILED DESCRIPTION:
OBJECTIVES

The proposed trial will randomize women and men with stage 0/I breast cancer scheduled for a lumpectomy, including excisional biopsy, ± sentinel node biopsy to one of three groups: 1) surgery with a local anesthetic, fentanyl, and HS before and during surgery (HS); 2) HS before surgery with usual care general anesthesia (HS-GA; total intravenous anesthesia rendering the patient unconscious with propofol infusion, airway instrumentation with a laryngeal mask airway or endotracheal tube, fentanyl, and local anesthetic); or 3) Usual care general anesthesia same as HS-GA group (GA). This project will allow further exploration of HS during surgery and to explore the biopsychosocial processes associated with analgesia and opioid use, anesthesia, and pain. We will test the hypotheses that HS during breast cancer surgery leads to reduced analgesia and opioid use, less pain and psychological stress, and faster recovery, as well as being more cost effective than GA or HS before surgery with GA.

Primary Objective:

To determine the efficacy of HS provided by a nurse anesthetist before and during surgery versus HS-GA or GA on reducing morphine equivalent daily dose (MEDD) from day of surgery through post-operative day (POD) 14.

Secondary Objectives:

* To determine the efficacy of HS with local anesthesia vs HS-GA or GA on reducing self-reported and objective pain, anxiety, nausea/vomiting, fatigue, and cognitive dysfunction.
* To evaluate group differences in costs. Using time and motion studies and methods of economic evaluation, we will test the hypothesis that HS before and during surgery will lead to less time spent in the OR and PACU, lower medication use, and less need for clinical staff engagement, leading to lower overall day of surgery-related costs.
* To explore psychosocial factors as moderators of the effects of the intervention and predictors of recovery. Baseline psychosocial factors including absorption, state and trait anxiety, intrusive thoughts, and discomfort intolerance, pain sensitivity, and expectations will moderate the effects of HS and predict outcomes over time.

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women;
2. Age 18 or older;
3. Diagnosed with stage 0/1 BCa;
4. Scheduled for a unilateral, segmental mastectomy, including excisional biopsy, ± SLND
5. Able to read, write and speak English or Spanish
6. Able to sign a written informed consent and be willing to follow protocol requirements.

Exclusion Criteria:

1. Extreme mobility issues that preclude participating in the study
2. Major thought disorders such as schizophrenia or uncontrolled bipolar disorder or PTSD
3. History of chronic opioid use
4. Current pain 2 or above on 0-10 scale
5. Co-mobilities such as uncontrollable diabetes or hypertension
6. Plastic surgery involvement for oncoplastic reconstruction
7. Have undergone chemotherapy for current breast cancer diagnosis
8. Surgery is likely greater than 3 hours
9. Patients with hearing loss that could preclude HS facilitation
10. Known allergy to propofol or other medications used during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Morphine Equivalent Daily Dose (MEDD) | through study completion; an average of 1 year.
  To determine the efficacy of HS provided by a nurse anesthetist before and during surgery versus HS-GA or GA on reducing morphine equivalent daily dose (MEDD) from day of surgery through post-operative day (POD) 14.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT05766891/ICF_000.pdf